CLINICAL TRIAL: NCT05083546
Title: Testing the Impact of a Combination of Dietary Supplements With Multimodal Effects on Longevity Mechanisms on Reducing Body Weight and Delaying Aging
Brief Title: Methylglyoxal (MGO) Lowering Cocktail to Reduce Appetite in Obese Individuals
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No funding
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-32631
Record Dates: First submitted 2021-07-26; First posted 2021-10-19 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Aging
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Double-Blinded, Randomized Control Trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be computer sequence-randomized to receive either oral daily dosing ofthe MGO cocktail or placebo. Both participants and study team members will be blinded to treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): MGO cocktail containing a combination of alpha-lipoic acid, nicotinamide, thiamine, pyridoxamine, and piperine
  Interventions: Drug: Gly-low
- Control (Placebo Comparator): sugar pill
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Gly-low — MGO cocktail containing a combination of alpha-lipoic acid, nicotinamide, thiamine, pyridoxamine, and piperine
  Arms: Intervention
Other: Placebo — sugar pill
  Arms: Control

SUMMARY:
Mechanisms that drive addiction to sugar rich foods are a major driving factor in the pathogenesis of obesity, which has become one of the most significant health care burdens. The molecular underpinnings of these hedonic mechanisms that drive addiction to sugar are poorly understood. The investigators demonstrated that methylglyoxal (MGO) derived Advanced Glycation Endproducts (AGEs) enhance food intake especially under a high sugar diet. The investigators identified a methylglyoxal (MGO) lowering cocktail, Gly-low, a combination of alpha-lipoic acid, nicotinamide, thiamine, pyridoxamine, and piperine that demonstrates a multimodal effect influencing many pathways related to aging including calorie restriction. Glycation lowering (Gly-low) treatment significantly reduces food intake and weight gain in the db/db mice that lack the leptin receptor. The investigators also extended the lifespan of C57BL/6 mice fed with these compounds starting when they were 24 months old. Based on these results, the investigators hypothesized that methylglyoxal (MGO) lowering cocktail of compounds can be given to adults with obesity, specified as body mass index (BMI) >27, to lower serum and urinary markers of insulin resistance, lower boy mass index (BMI), and lower food intake.

DETAILED DESCRIPTION:
The aging population in the United States of America and around the world is expected to put enormous pressure on the medical system and thus aging remains the biggest challenge for biomedicine. The current approaches to slow aging or age-related diseases rely on targeting specific pathways for each indication, whereas the cause of aging is multifactorial. Hence, developing drugs that can function in a multimodal fashion to engage multiple pathways involved in aging is likely to be a much more effective approach.

Previous studies have demonstrated that combining mutations in the insulin and tOR (target of rapamycin) pathway can result in a nearly five-fold extension in lifespan. This study proposes to achieve similar effects pharmacologically. A compound mix has been identified utilizing glycation lowering (Gly-low) compounds that alter multiple key pathways involved in aging including the reduction of calorie intake, Nicotinamide adenine dinucleotide (NAD) metabolism, inflammation, glycation stress and increased fat burning. Preliminary findings that have shown significant increases in survival of normal and diabetic mice models fed with Gly-low confirms the efficacy of multimodal benefits of Glycation lowering (Gly-low) compounds. Glycation lowering (Gly-low) compounds were chosen based on their ability to protect neurons against glycation stress and consist of 5 compounds that have been designated GRAS (generally regarded as safe) by the Food and Drug Administration (FDA). Based on these results, the investigators hypothesize that methylglyoxal (MGO) lowering cocktail of compounds can be given to adults with obesity, specified as body mass index body mass index (BMI) >27, to lower serum and urinary markers of insulin resistance, lower body mass index (BMI), and lower food intake. Successful completion of this innovative project will result in a cocktail of compounds that can complement ongoing treatments to reduce obesity and enhance the health and slow age-related diseases.

This is a single center, double-blind, placebo-controlled, randomized trial. 100 subjects will be recruited between the ages of 50 and 70 yrs with a body mass index (BMI)>27. The participant will take 3 Gly-low supplements in pill form orally by mouth once in the morning. Baseline measurements in body mass index (BMI) (height and weight), waist circumference, food intake and dietary behavior (by questionnaire), urine, and serum will be obtained. Body mass index (BMI) will be measured every 12 weeks. The primary endpoints will be measures of physical frailty, based on performance and a clinical frailty index, and cognitive performance based on a cognitive impairment questionnaire, including memory, will be measured after 6 months and 12 months. Urine and serum will be analyzed every 12 weeks for various aging and metabolic markers. Patients will also be monitored for side effects or other compound related issues.

Screening data will be reviewed to determine subject eligibility. Subjects who meet all inclusion criteria and none of the exclusion criteria will be entered into the study.

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI >27) individuals

Exclusion Criteria:

* must be older than 50 years of age or older

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in body mass index (BMI) from baseline to 1 year | baseline and one year
  Body Mass Index (BMI) is a calculated from a person's weight in kilograms divided by the square of height in meters.
Change in frailty from baseline to 1 year | baseline and 1 year
  Frailty will be assessed and measured using a questionnaire-based method as well as analyzing the physical performance of the subject in clinic. The Clinical Frailty Scale (CFS) is a judgement-based frailty tool that evaluates specific domains including comorbidity, function, and cognition to generate a frailty score ranging from 1 (very fit) to 9 (terminally ill).
Change of cognition from baseline to 1 year | baseline to 1 year
  Cognition will be assessed and measured using a questionnaire-based method. The Clinical Frailty Scale (CFS) is a judgement-based frailty tool that evaluates specific domains including comorbidity, function, and cognition to generate a frailty score ranging from 1 (very fit) to 9 (terminally ill).

SECONDARY OUTCOMES:
Blood Marker Glucose for Aging and Insulin Resistance | baseline to 1 year
  Blood samples will be collected and analyzed over the course of the study to measure the blood marker glucose in mmol/L associated with aging and insulin resistance.

OTHER OUTCOMES:
Blood Marker Insulin for Aging and Insulin Resistance | baseline to 1 year
  Blood samples will be collected and analyzed over the course of the study to measure the blood marker insulin in ulU/mL associated with aging and insulin resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Stoller, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.